CLINICAL TRIAL: NCT02662881
Title: Post-Market Data Collection for Biologically Assisted Core Decompression of the Femoral Head Using the PerFuse Instrument and BioCUE
Brief Title: Biologically Assisted Core Decompression of the Femoral Head Using the PerFuse Instrument and BioCUE
Acronym: REGP-44-00
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: BBIO.CR.BIOAVN.002.15
Record Dates: First submitted 2016-01-18; First posted 2016-01-26 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Avascular Necrosis of the Femoral Head
MeSH Terms: conditions — Femur Head Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PerFuse Percutaneous Decompression System — Core decompression with PerFuse
Device: BioCUE Platelet Concentration System — PRP injection through the PerFuse cannula into core decompression site

SUMMARY:
This study will evaluate the performance of biologically assisted core decompression with the PerFuse instrument and BioCUE in patients with bone lesions in the femoral head. The study will explore the potential impact of patient demographics and baseline characteristics on post-operative outcomes.

DETAILED DESCRIPTION:
This study will evaluate the performance of biologically assisted core decompression with the PerFuse instrument and BioCUE in patients with bone lesions in the femoral head. The study will explore the potential impact of patient demographics and baseline characteristics on post-operative outcomes. The study will evaluate change in Harris Hip Score (HHS) at 12 months after treatment. The change in AVN lesion size will also be measured at 12 months after index treatment via MRI. Change in quality of life and pain measures will be measured at each follow-up. Adverse events will also be recorded throughout the study.

This study will follow patients for 5 years after initial treatment.

Data will be recorded in a online database that will be entered by the site or patient, depending on the report form. This database includes data checks to compare entered data against predefined rules for range.

A risk-based monitoring plan will be put in place for source data verification.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with the study procedures
* Signed informed consent
* Untreated unilateral or bilateral bone lesion(s) of the femoral head associated with AVN in need of biologically assisted core decompression. Note:If bilateral untreated bone lesions of the femoral head associated with AVN,both hips eligible and willing to undergo study treatment and follow-up
* ≥ 3 months after arthroplasty (e.g., total, hemi) in the contralateral hip

Exclusion Criteria:

* Pregnant or lactating
* Participating in another device or drug study
* ARCO stage ≥ III
* Unable to undergo MRI of the study hip(s)
* Active, local or systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with untreated unilateral or bilateral bone lesion(s) of the femoral head associated with AVN in need of biologically assisted core decompression.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score | 12 month
  Percentage of patients achieving clinical success at 12 month follow up, being defined as a 20 point increase in the Harris Hip Score from baseline

SECONDARY OUTCOMES:
Incidence of invasive non-study procedures in the hip | 5 years (all time points)
  Number of hip requiring an non-study invasive procedure
Second procedure | 5 years (all time points)
  Number of patients receiving a second study procedure
Hips with no lesion size change | 12 months
  Number of hips with no change or reduction in lesion size
Adverse Events | 5 years (all time points)
  Number of adverse events
Harris Hip Score | 5 years (all time points)
  number of patients with "Good" or "Excellent" scores
EQ-5D-3L | 5 years (all time points)
  Change in European Quality of Life 5 Dimensions 3 Levels score
NRS Pain | 5 years (all time points)
  Change in Numeric Rating Scale for Pain score

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Travers, MD, Principal Investigator — Trustees of the University of Pennsylvania; Cecilia Pasucal-Garrido, MD, Principal Investigator — Washington University School of Medicine; Joseph Schwab, MD, Principal Investigator — Medical College of Wisconsin; Nicolas Piuzzi, MD, Principal Investigator — The Cleveland Clinic
Locations (4):
- United States (4):
  - Washington University in St. Louis, St Louis, Missouri
  - Cleveland Clinic Foundation - Orthopaedic and Rheumatologic Institute, Cleveland, Ohio
  - University of Pennsylvania/ Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Medical College Of Wisconsin, Milwaukee, Wisconsin